CLINICAL TRIAL: NCT03289832
Title: Effect of Orally Delivered Phytochemicals, Alone, and in Combination, on Aging and Inflammation-Related Effects in the Skin
Brief Title: Effect of Orally Delivered Phytochemicals on Aging and Inflammation in the Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00117754
Record Dates: First submitted 2017-08-10; First posted 2017-09-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Healthy Adults
Keywords: Sulforaphane; Curcumin; Crucera-SGS; Meriva-SF; Skin; erythema; UV; Sunburn; Inflammation; Redness; ultra-violet; sunlight
MeSH Terms: conditions — Erythema; Sunburn; Inflammation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Crucera-SGS® (Active Comparator): Drug: Subjects will follow a cruciferous vegetable-free diet and will first undergo a 10 day nonintervention phase. For the second phase they will be instructed to maintain a non-cruciferous diet and to ingest daily for 10 days, Crucera-SGS® as a source of glucoraphanin which is converted to sulforaphane; 9 capsules (450 mg or 1.03 mmol GR) per day.
  On the 7th day of each phase, they will be asked to fast overnight, come in to the clinic, provide urine and blood, and receive a dose 2-times their M.E.D. at up to 5 sites on the upper buttocks. Following the first and third days of chromometer readings, 2 biopsies will be taken from the upper buttocks for a total of 8 skin-punch biopsies per individual.
  Interventions: Dietary Supplement: Crucera-SGS
- Meriva 500-SF® (Active Comparator): Drug: Subjects will follow a cruciferous vegetable-free diet and will first undergo a 10 day nonintervention phase. For the second phase they will be instructed to maintain a non-cruciferous diet and to ingest daily for 10 days, Meriva 500-SF® as a source of curcumin; 2 capsules (1000 mg or 2.72 mmol total curcuminoids) per day.
  On the 7th day of each phase, they will be asked to fast overnight, come in to the clinic, provide urine and blood, and receive a dose 2-times their M.E.D. at up to 5 sites on the upper buttocks. Following the first and third day of chromometer readings, 2 biopsies will be taken from the upper buttocks, for a total of 8 skin-punch biopsies per individual.
  Interventions: Dietary Supplement: Meriva 500-SF
- Crucera-SGS® and Meriva 500-SF® (Active Comparator): Drug: Subjects will follow a cruciferous vegetable-free diet and will first undergo a 10 day nonintervention phase. For the second phase they will be instructed to maintain a cruciferous vegetable-free diet and to ingest daily for 10 days, Crucera-SGS® as a source of glucoraphanin which is converted to sulforaphane; 9 capsules (450 mg or 1.03 mmol GR) and Meriva 500-SF® as a source of curcumin; 2 capsules (1000 mg or 2.72 mmol total curcuminoids) per day.
  On the 7th day of each phase, they will be asked to fast overnight, come in to the clinic, provide urine and blood, and receive a dose 2-times their M.E.D. at up to 5 sites on the upper buttocks. Following the first and third day of chromometer readings, 2 biopsies will be taken from the upper buttocks for a total of 8 skin-punch biopsies per individual.
  Interventions: Dietary Supplement: Crucera-SGS; Dietary Supplement: Meriva 500-SF

INTERVENTIONS:
Dietary Supplement: Crucera-SGS — Crucera-SGS is a commercially available dietary supplement. The active ingredient is glucoraphanin, a phytochemical from broccoli and it is prepared as a simple extract of broccoli seeds. Glucoraphanin is converted to sulforaphane by bacteria in the human intestines. Crucera-SGS is formulated by Thorne Research Inc. into gel-caps that make it much more convenient to deliver than having subjects eat broccoli every day.
  Arms: Crucera-SGS®; Crucera-SGS® and Meriva 500-SF®
Dietary Supplement: Meriva 500-SF — Meriva-SF is a commercially available dietary supplement. The active ingredient is curcumin, a phytochemical from the spice, turmeric, and it is prepared as a simple extract of this plant, formulated with lipids which aid in its absorption and metabolism. Meriva-SF is formulated by Thorne Research Inc. into gel-caps that make it much more convenient to deliver than having subjects eat turmeric powder every day.
  Arms: Crucera-SGS® and Meriva 500-SF®; Meriva 500-SF®

SUMMARY:
The objective is to determine, in a small number of participants, the protective effects of UV-induced skin erythema (reddening or "sunburn") following oral administration of sulforaphane, curcumin, or a combination of the two plant (diet)-based supplements. The investigators will be using the over-the-counter nutritional supplements Crucera-SGS and Meriva-SF to deliver the biologically stable sulforaphane precursor and a highly bioavailable formulation of curcumin. Volunteers will be challenged with UV irradiation at 2-times the minimum erythematous dose (M.E.D.) on discrete 2 cm diameter circles on the upper buttocks. Skin redness will be monitored daily using a chromometer. Biomarkers will then be evaluated in blood, urine, and skin biopsies.

DETAILED DESCRIPTION:
Oral sulforaphane (SF) delivery results in systemic protection of a wide variety of organ systems which The investigators hypothesize will also include the skin, based on animal studies and preliminary evidence in human volunteers. Since The investigators have only previously evaluated the ability of topical sulforaphane application to protect skin from UV-induced erythema, the next logical step is to evaluate the ability of oral delivery to affect the skin of healthy human volunteers. Curcumin is also a potent anti-inflammatory that acts upon different biochemical pathways from SF, and it is an antioxidant. It was discovered over a century ago, it has been the subject of well over a hundred clinical studies, and it has been an ingredient in common foods eaten by millions of people, for centuries. Before and after consumption of each of these common food ingredients, The investigators will: (a) measure the Phase 2 cytoprotective response in human skin, (b) determine whether it leads to reduced UV-induced erythema (reduced inflammation), (c) evaluate changes in age-related markers such as dermal elasticity, keratin and collagen levels, (d) measure advanced glycation end-products (AGEs) in the serum, as biomarkers of systemic (including the skin) reduction in AGE levels, and (e) measure the levels of these biomarkers in skin punch biopsies. The investigators will also evaluate the effects of combined oral SF and curcumin. The investigators anticipate that there may be a true synergistic response between SF and curcumin, and the experiments designed herein are designed to show that synergy, if it exists.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old, healthy
* Willingness to avoid sun exposure to study site
* Willingness to adhere to cruciferous vegetable-free diet

Exclusion Criteria:

* Use of photosensitizing medications
* Use of medications that cause skin flushing
* Use of anticoagulants/antiplatelet therapies
* Allergies to anesthetic agents
* Use of systemic retinoids or steroids (excluding female contraceptives and levothyroxin)
* Topical retinoids or steroids at study sites
* Antibiotic use
* Current students of the Principal Investigator
* Procedures performed at the study sites
* Smokers/tobacco users

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
Change in Erythema 1 Day After UV Exposure | On day 8 of intervention
  Brief ultraviolet (UV) exposure on small circular spots on the skin will produce erythema (reddening), to be measured with a chromameter and photographed in the days following UV exposure, both before and after subjects have ingested study supplement (Crucera SGS, Meriva 500-SF, or both), daily, for a week. These measures will be compared to erythema in the skin of the same individuals following UV exposure, but WITHOUT having ingested these supplements.
Change in Erythema 2 Days After UV Exposure | On day 9 of intervention
  Brief ultraviolet (UV) exposure on small circular spots on the skin will produce erythema (reddening), to be measured with a chromameter and photographed in the days following UV exposure, both before and after subjects have ingested study supplement (Crucera SGS, Meriva 500-SF, or both), daily, for a week. These measures will be compared to erythema in the skin of the same individuals following UV exposure, but WITHOUT having ingested these supplements.
Change in Erythema 3 Days After UV Exposure | On day 10 of intervention
  Brief ultraviolet (UV) exposure on small circular spots on the skin will produce erythema (reddening), to be measured with a chromameter and photographed in the days following UV exposure, both before and after subjects have ingested study supplement (Crucera SGS, Meriva 500-SF, or both), daily, for a week. These measures will be compared to erythema in the skin of the same individuals following UV exposure, but WITHOUT having ingested these supplements.

SECONDARY OUTCOMES:
Bioavailability of Supplement Metabolites in bodily fluids | Day 7 of each phase of intervention
  Metabolites of both sulforaphane and curcumin will be measured in blood and/or urine samples. Curcumin is rapidly conjugated to glucuronides and sulfates, which will be enzymatically degraded prior to measurement. Glucosinolates are metabolized to sulforaphane which is in turn metabolized to compounds collectively called dithiocarbamates. All of these can be readily measured using the cyclocondensation assay which reacts with all of the dithiocarbamates to produce a chromogenic compound with a very high molar extinction coefficient that is measured spectrophotometrically. Comparing levels before and after intervention will allow inferences to be made about bioavailability.
Change in metabolomic profile | Day 7 of each phase of the intervention
  Blood samples taken before- and after- the intervention in each of the treated arms will be assessed for an extensive spectrum of small-molecule metabolites. Assessment will be by Mass Spectroscopy, in what is known as an untargeted metabolomic screen. Statistically-assisted exploration of this data-set is expected to yield insight into the metabolic pathways that are up- and down- regulated (boosted or supressed [inhibited]) as a result of treatment with these supplements.
Change in tissue-based RNA biomarkers of inflammation | Up to day 8 of intervention
  Biomarkers of inflammation will be measured in skin-punch biopsies. Biopsy measures will reflect inflammation at the site of reddening (e.g. sunburn). A limited [by tissue availability] number of assessments will be made by real time PCR.
Change in tissue-based protein biomarkers of inflammation | Up to day 10 of intervention
  Biomarkers of inflammation will be measured in skin-punch biopsies. Biopsy measures will reflect inflammation at the site of reddening (e.g. sunburn). A limited [by tissue availability] number of assessments will be made by ELISA, protein blotting and immunohistochemistry.
Change in blood-based biomarkers of inflammation | Day 7 of each phase of the intervention
  Biomarkers of inflammation will be measured in blood, and will reflect systemic (whole body) effects that are not likely to be large. An extended panel of inflammatory cytokines and cytoprotective enzymes may be evaluated. Assessments will be by real time PCR, ELISA, and protein blotting.
Change in urine-based biomarkers of inflammation | Day 7 of each phase of the intervention
  Biomarkers of inflammation will be measured in urine, and will reflect systemic (whole body) cumulative effects that are not likely to be large. An limited panel of inflammatory cytokines and cytoprotective enzymes may be evaluated. Assessments will be by real time PCR, ELISA, and protein blotting.
Change in RNA markers of aging and protection from UV damage | Up to day 8 of intervention
  Skin-punch biopsies will be evaluated for markers of an up-regulated cytoprotective response including protection from photooxidation damage, and biomarkers of aging that may include advanced glycation end-products (AGE), skin elasticity, keratins, and collagens. Assessments will be by real time PCR.
Change in protein and small-molecule markers of aging and protection from UV damage | Up to day 10 of intervention
  Skin-punch biopsies will also be evaluated for markers of an up-regulated cytoprotective response including protection from photooxidation damage, and biomarkers of aging that may include advanced glycation end-products (AGE), skin elasticity, keratins, and collagens. Assessments will be by ELISA, protein blotting and immunohistochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Jed W Fahey, ScD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No